CLINICAL TRIAL: NCT03343743
Title: Changes in Renal Papillary Density After Hydration Therapy in Calcium Stone Formers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6118/13
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydration (Other): Patients were instructed to drink at least 2 L/day of a hypotonic, oligomineral water low in sodium and minerals (fixed residue at 180°C <200 mg/L) for at least 12 months
  Interventions: Other: Oligomineral water

INTERVENTIONS:
Other: Oligomineral water — Patients were instructed to drink at least 2 L/day of a hypotonic, oligomineral water low in sodium and minerals (fixed residue at 180°C <200 mg/L) for at least 12 months

SUMMARY:
Patients with recurrent calcium oxalate stones undergoing endourological procedures for renal stones at our institution from June 2013 to June 2014 were considered eligible for enrolment. Enrolled patients underwent a baseline unenhanced CT scan before the urological procedure; after endoscopic removal of their stones, the patients were instructed to drink at least 2 L/day of a hypotonic, oligomineral water low in sodium and minerals (fixed residue at 180°C <200 mg/L) for at least 12 months. Finally, the patients underwent a follow-up unenhanced CT scan during hydration regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing endourological procedures for renal stones
* Recurrent stone disease
* Calcium oxalate stones (>50% of the stone made of calcium oxalate)

Exclusion Criteria:

* Systemic conditions causing stones (hyperparathyroidism, intestinal malabsorption, renal tubular acidosis)
* Non-calcium oxalate stones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Changes in renal papillary density | At baseline and after 12 months
  Renal papillary density measured with unenhanced CT scan

REFERENCES:
- [Derived] Ferraro PM, Vittori M, Macis G, D'Addessi A, Lombardi G, Palmisano C, Gervasoni J, Primiano A, Bassi PF, Gambaro G. Changes in renal papillary density after hydration therapy in calcium stone formers. BMC Urol. 2018 Nov 12;18(1):101. doi: 10.1186/s12894-018-0415-7. PMID 30419887